CLINICAL TRIAL: NCT02020720
Title: Evaluating the Impact of 18F-DOPA-PET on Neurosurgical Planning for Gliomas
Brief Title: 18F-DOPA-PET in Planning Surgery in Patients With Gliomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1373; P50CA108961 (NIH); R01CA178200 (NIH); NCI-2013-02373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1373 (Other: Mayo Clinic); 13-005102 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Malignant Glioma; Recurrent Brain Neoplasm
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Biopsy; fluorodopa F 18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-DOPA-PET) (Experimental): Within 1 week of biopsy or resection, patients undergo 18F-DOPA PET/CT scan and pMRI and DTI at baseline. Patients then undergo stereotactic craniotomy or image-guided biopsy.
  Interventions: Procedure: Biopsy; Procedure: Computed Tomography; Procedure: Diffusion Weighted Imaging; Drug: Fluorine F 18 Fluorodopa; Other: Laboratory Biomarker Analysis; Procedure: Perfusion Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biopsy — Undergo image-guided biopsy
  Other Names: Bx
Procedure: Computed Tomography — Undergo 18F-DOPA-PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Diffusion Weighted Imaging — Undergo DTI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Drug: Fluorine F 18 Fluorodopa — Undergo 18F-DOPA-PET/CT
  Other Names: 18F-FDOPA
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Perfusion Magnetic Resonance Imaging — Undergo pMRI
  Other Names: magnetic resonance perfusion imaging
Procedure: Positron Emission Tomography — Undergo 18F-DOPA-PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Therapeutic Conventional Surgery — Undergo stereotactic craniotomy

SUMMARY:
This pilot clinical trial studies fluorine F 18 fluorodopa (18F-DOPA)-positron emission tomography (PET) in planning surgery in patients with gliomas. New imaging procedures, such as 18F-DOPA-PET scan, may help find gliomas and may help in planning surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Accurately define a standardized 18F-DOPA PET tumor/normal tissue (T/N) threshold to delineate high grade gliomas (HGG) from low grade gliomas (LGG).

SECONDARY OBJECTIVES:

I. Determine correlation between 18F-DOPA PET activity, magnetic resonance imaging (MRI) contrast enhancement and high- or low-grade glioma biopsies.

II. Compare grade from maximum 18F-DOPA uptake samples for all resection patients against the final diagnostic grade, based on the highest grade component from all stereotactic and non-stereotactic samples acquired for open resection patients.

III. Compare volume differences between 18F-DOPA PET activity, MRI contrast enhancement, perfusion MRI (pMRI), and diffusion tensor imaging (DTI) for neurosurgical planning.

IV. Assess the time to progression for patients receiving resections and biopsies only.

TERTIARY OBJECTIVES:

I. Compare histopathology correlations with 18F-DOPA PET against correlations with perfusion MR imaging for accurate identification of the highest grade/highest density disease.

II. Compare histopathology correlations with 18F-DOPA PET against correlations with diffusion tensor imaging information for accurate identification of tumor extent.

III. Compare neurosurgical resection extent volume delineation with and without 18F-FDOPA-PET metabolic imaging information to determine role of metabolic imaging in neurosurgical resection planning.

OUTLINE:

Within 1 week of biopsy or resection, patients undergo 18F-DOPA PET/computed tomography (CT) scan and pMRI and DTI at baseline. Patients then undergo stereotactic craniotomy or image-guided biopsy.

After completion of study treatment, patients are followed up yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* MRI findings compatible with newly diagnosed or recurrent high- or low-grade malignant glioma
* Planned craniotomy and resection or biopsy
* Willing to sign release of information for any radiation and/or follow-up records
* Provide informed written consent if >= 18 years; if < 18 years, provide informed written assent and parent or legal guardian provide informed written consent
* Ability to provide tissue for mandatory correlative research component

Exclusion Criteria:

* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure)
* Unable to undergo an 18F-DOPA PET scan (e.g. Parkinson's disease, taking anti-dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists; NOTE: other potentially interfering drugs: amoxapine, amphetamine, benztropine, buproprion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, selegiline, paroxetine, citalopram, and sertraline; if a patient is on any of these drugs, list which ones on the on-study form
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Ratios of maximum tumor standardized uptake value (SUVmax) normalized to mean SUV (SUVmean) of T/N | Up to 1 year
  To determine the optimal PET threshold for distinguishing HGG from LGG brain tissue, receiver operating characteristic (ROC) analysis and the Youden's index (sum of the sensitivity and specificity - 1) will be used. The Youden's index will be calculated for each possible T/N threshold. The final ROC area under the curve (AUC) value and confidence intervals will be estimated using ROC analysis methods for clustered continuous data as described by Obychowski.

SECONDARY OUTCOMES:
Differences in volumes generated from biopsy-validated thresholds evaluated by 18F-DOPA-PET, pMRI, and DTI | Up to 5 years
  Paired t-test statistical analysis will be performed to determine if any differences exist and the level of statistical significance between volumes.
Histologic grade of the specimen defined as HGG, LGG, or non-malignant brain tissue | Up to 5 years
  The relationship between these T/N values, MRI contrast enhancement values, and the histologic grade of the specimen (HGG, LGG, or non-malignant brain tissue) will be determined using multivariate linear regression. These models will also include as appropriate the specimen cellularity and necrosis values.
MRI contrast enhancement values | Up to 5 years
  The relationship between these T/N values, MRI contrast enhancement values, and the histologic grade of the specimen (HGG, LGG, or non-malignant brain tissue) will be determined using multivariate linear regression. These models will also include as appropriate the specimen cellularity and necrosis values.
Progression free survival | The time from study entry to progression, assessed up to 5 years
Proportion of patients whose maximum 18F-DOPA uptake samples are in agreement with the final diagnostic grade | Up to 5 years
  Associated confidence intervals will be estimated based on dividing the number of patients whose samples agree by the total number of patients.

OTHER OUTCOMES:
Accurate identification of the highest grade/highest density disease | Up to 5 years
  Paired t-test statistical analysis will be used to evaluate differences in volumes identified using biopsy-validated thresholds as highly aggressive disease comparing 18F-DOPA uptake and relative cerebral blood volume from pMRI.
Accurate identification of tumor extent | Up to 5 years
  Paired t-test statistical analysis will be used to evaluate differences in volumes identified using biopsy-validated thresholds as disease extent comparing 18F-DOPA PET and diffusion maps from DTI.
Role of metabolic imaging in neurosurgical resection planning | Up to 5 years
  Paired t-test analysis will be performed to determine the level of statistical significance between conventional MRI only and PET + MRI volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, M.D., Principal Investigator — Mayo Clinic in Rochester; Debra H. Brinkmann, Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials